CLINICAL TRIAL: NCT01617876
Title: A Prospective Study on the Accuracy of Enhanced Magnifying Endoscopy for Differential Diagnosis of Small Focal Gastric Lesions Identified With White-light Endoscopy
Brief Title: Enhanced Magnifying Endoscopy for Diagnosis of Early Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Xinghua Lu, Chairman of Beijing Institute of Digestive Endoscopy of Chinese Medical Association, Peking Union Medical College Hospital
Other Study IDs: LXH-EGC-1; 200902002 (Other Grant/Funding Number: Ministry of Health of China)
Record Dates: First submitted 2012-06-09; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; early gastric cancer; magnifying endoscopy; narrow band imaging; acetic acid; indigocarmine
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy of gastric lesions
Oversight: Data Monitoring Committee: No

SUMMARY:
When performing screening endoscopy, small focal gastric lesions are frequently encountered. Novel techniques in endoscopy, such as magnifying endoscopy (ME) with narrow-band imaging (NBI) and chromoendoscopy with acetic acid-indigocarmine mixture (AIM), are developing to enhance images of gastrointestinal tumor. Furthermore, observation of the microstructures of gastric mucosa by ME, including microvascular pattern and microsurface pattern, has been proposed in the recognition of early gastric cancer (EGC).

This study is based on the hypothesis as follow:

1. The microvascular structure could be clearly observed with magnifying endoscopy enhanced by narrow-band imaging (ME-NBI).
2. The microsurface architecture could be clearly observed with magnifying endoscopy enhanced by acetic acid-indigocarmine mixture (ME-AIM).
3. Enhanced ME (combining ME-NBI and ME-AIM), as compared to white-light endoscopy (WLE), has higher sensitivity and specificity for the differential diagnosing small focal gastric lesions.

DETAILED DESCRIPTION:
Patients who received surveillance endoscopy for EGC using a zoom endoscope were eligible for inclusion. WLE without magnification was performed first in eligible patients. Based on an assessment of the shape (such as flat, depressed or elevated) and color (pale or reddened), small focal gastric lesions were identified and included for evaluation by experienced endoscopists. When such a lesion was detected during non-magnifying observation with WLE, the mode was then changed to ME-NBI for observation of microvascular pattern and ME-AIM for observation of microsurface pattern subsequently. All endoscopic images of the whole procedure were recorded in digital filing system for later evaluation. To avoid possible selection bias and to maintain the quality of the study, all images of each endoscopic modality (including WLE, ME-NBI, ME-AIM), which were arranged randomly on one slide and displayed independently of the images of other endoscopic modality, were evaluated by 4 skilled endoscopists, who were not access to the clinical and pathological data. The general consensus was established for an assessment of each lesion. Two forceps biopsy specimens were taken from each lesion and pathological diagnosis were used as the criterion standard for cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients, in which small focal gastric lesions were identified with conventional WLE, were enrolled in this study. Before being enrolled, all patients provided written informed consent.

Exclusion Criteria:

* Patients who cannot undergo gastroscopies due to unsuitable conditions
* Referred patients with a history of having being diagnosed as gastric cancer
* Patients with a personal history of gastric surgery
* Patients who cannot provide informed consent
* Patients with advanced gastric cancer

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received surveillance endoscopy for EGC using a zoom endoscope were eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of enhanced ME (combining ME-NBI and ME-AIM) | 1 week
  Enhanced ME diagnosis was made subsequent to endoscopy procedure and reviewed in a week when confirmed histopathologic diagnosis was out for comparison. Percentage of sensitivity, specificity, positive predictive value and negative predictive value of enhanced ME diagnosis compared with histopathology diagnosis were measured.

SECONDARY OUTCOMES:
Diagnostic accuracy of WLE | 1 week
  WLE diagnosis was made subsequent to endoscopy procedure and reviewed in a week when confirmed histopathologic diagnosis was out for comparison. Percentage of sensitivity, specificity, positive predictive value and negative predictive value of WLE diagnosis compared with histopathology diagnosis were measured.
The relationships between the microvascular patterns and the histopathological findings | 1 week
  The microvascular pattern of each lesion was evaluated subsequent to endoscopy procedure and reviewed in a week when confirmed histopathologic diagnosis was out for comparison. Percentage of distribution of different microvascular patterns compared with histopathology diagnosis was measured.
The relationships between the microsurface patterns and the histopathological findings | 1 week
  The microsurface pattern of each lesion was evaluated subsequent to endoscopy procedure and reviewed in a week when confirmed histopathologic diagnosis was out for comparison. Percentage of distribution of different microsurface patterns compared with histopathology diagnosis was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Lu, Dr, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Gastroenterology, Peking Union Medical College Hospital, Beijing, China